CLINICAL TRIAL: NCT03515863
Title: Natural History and Genetic Risk Factors of Thyroid Associated Ophthalmopathy (TAO)
Brief Title: Natural History and Risk Factors of TAO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Clinical investigator, Sun Yat-sen University
Other Study IDs: 2017KYPJ123
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Thyroid Associated Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grave's disease with TAO: Patients with Grave's disease and TAO
  Interventions: Genetic: DNA extraction and genetic characterization; Device: Orbit MRI examination; Other: Collection of life style data
- Grave's disease without TAO: Patients with Grave's disease but without TAO
  Interventions: Genetic: DNA extraction and genetic characterization; Device: Orbit MRI examination; Other: Collection of life style data

INTERVENTIONS:
Genetic: DNA extraction and genetic characterization — Collection of blood samples for DNA extraction and genetic characterization using whole-genome sequencing, and for identification of cellular biomarkers using transcriptomics and mass cytometry.
Device: Orbit MRI examination — Orbit MRI examination is performed to confirm the diagnosis of TAO
Other: Collection of life style data — Collection of life style data using quality of life questionnaire

SUMMARY:
The aim of this study is to complete the identification of genetic factors predisposing to thyroid associated ophthalmopathy (TAO) by constituting a cohort of 400 Grave's patients with or without ocular signs.

DETAILED DESCRIPTION:
Graves' disease (GD) is a common autoimmune condition, and its ocular condition is known as thyroid-associated ophthalmopathy (TAO). There is considerable evidence that both genetic and environmental factors are involved in the development of TAO. We conduct a study of 400 Grave's patients, with or without TAO, and obtain the following data: genetic tests, ocular imaging and life style information. Genetic tests are obtained by collection of blood samples for DNA extraction, whole-genome sequencing, and identification of cellular biomarkers, using transcriptomics and mass cytometry. Ocular imaging data are collected from Orbit MRI examination. Life style data are collected using a standardized questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of Grave's disease with the history of more than 1 years
2. Informed consent signed by a patient or legal guardian, or having the ability to comply with study assessments for the full duration of the study

Exclusion Criteria:

1. Pregnancy (positive test) or lactation
2. Participating in another simultaneous medical investigation or clinical trial within 3 months
3. Having received cellular therapy
4. With a history of psychotropic drugs abuse
5. With a history of mental disorder
6. With a history of malignant tumor
7. Any medical or social condition that in the judgment of the investigator would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TAO Patients:
  Patients who are diagnosed as Grave's disease and TAO are enrolled into the study from 2 clinical centers. This diagnosis is made according to classical criteria of TAO, including thyroid function testing, ocular examination and orbit MRI examination.
  Control:
  Patients who are diagnosed as Grave's disease but without ocular signs are enrolled into the study from 2 clinical centers. This diagnosis of Grave's disease is made according to classical criteria including thyroid function testing. Ocular signs are excluded by routine ocular examination and orbit MRI examination.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-05-09 (Estimated); Study Completion 2022-05-09 (Estimated)

PRIMARY OUTCOMES:
Genetic risk factors of TAO predisposition | 1 year
  Genetic risk factors of TAO are identified by pathogenic gene screening using the whole-genome sequencing of peripheral blood cells.

SECONDARY OUTCOMES:
Cellular biomarkers for risk of TAO | 1 year
  Cellular biomarkers for risk of TAO are identified by transcriptomics and mass cytometry

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - the First People's Hospital of Zhaoqing, Zhaoqing